CLINICAL TRIAL: NCT06554704
Title: Autonomic Nervous System Dysregulation in People With Chronic Neck Pain - Indicated by Heart Rate Variability
Brief Title: Autonomic Nervous System Dysregulation in People With Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: NYCU113077AE
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2024-07

CONDITIONS: Chronic Neck Pain; Autonomic Nervous System
Keywords: Heart rate variability; Isometric hand-grip test; Posture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic neck pain: Individuals with non-specific chronic neck pain
  Interventions: Behavioral: Isometric hand grip test
- Healthy control: Individuals without non-specific chronic neck pain
  Interventions: Behavioral: Isometric hand grip test

INTERVENTIONS:
Behavioral: Isometric hand grip test — The five-minute heart rate variability and respiration rate will be measured for each condition including resting in supine, sitting and standing position, as well as the isometric hand grip test in supine, sitting and standing position.

SUMMARY:
The goal of this observational study is to investigate heart rate variability in different positions and in response to isometric hand-grip test in people with non-specific chronic neck pain as compared with healthy controls. The main questions it aims to answer are:

* Do the heart rate variability indices differ between people with non-specific chronic neck pain and healthy controls in supine sitting and standing positions?
* Do the heart rate variability indices differ between people with non-specific chronic neck pain and healthy controls when challenged by the isometric hand-grip test?

DETAILED DESCRIPTION:
Background: Chronic neck pain (CNP) is a common symptom that affects the neck region with persistent or recurrent pain for more than 3 months. Ninety percent of people experience CNP is non-specific, meaning the underlying cause is not clear or specific. CNP is associated with risk factors that potentially induce sustained physiological responses. The autonomic nervous system (ANS) is responsible for controlling physiological functions and is required to adaptively respond to physical and mental stress. The risk factors may lead to ANS dysregulation and decrease capacity to cope with sensory and emotional stress. The ANS regulation can be measured through the assessment of heart rate variability (HRV). However, limited number of studies have documented the ANS dysregulation in people with CNP. The aim of present study is to investigate HRV in different positions and in response to isometric hand-grip (IHG) test in people with non-specific CNP as compared with healthy controls (HC).

Methods: This is an observational cross-sectional study. Twenty-eight participants with non-specific CNP and 28 age- and gender-matched HC will be recruited. The 5-min HRV and respiration rate will be measured for each condition including resting in supine, sitting and standing position, as well as the IHG test in supine, sitting and standing position. The 3-lead electrocardiography (ECG) data will be collected and analyzed for HRV indices, including time domain (mean R-R interval, standard deviation of the normal-to-normal interval and root mean square successive difference) and frequency domain (low frequency (LF), high frequency (HF) and LF/HF ratio). Statistical analysis: Descriptive data are presented as mean with standard deviation or frequency. Group differences in subject characteristics are analyzed using independent t-test or Chi-square test. Two-way mixed analyses of covariance (ANCOVAs) are used to assess HRV indices between groups and conditions with Tukey post hoc analysis. The maximal voluntary contraction of IHG test, pain intensity indicated by numeric rating scale and respiratory rate will be used as covariates. The significant level is set at p < 0.05.

ELIGIBILITY:
Chronic neck pain inclusion criteria:

* Chronic pain (persistent or recurrent pain >90 days)
* Non-specific chronic neck pain and non-irradiated to the upper limbs (Superior nuchal line ~ scapular spine ~ acromion)

Chronic neck pain & healthy control inclusion criteria:

* Age- and gender- matched (age: 20~59 y/o)
* BMI between 18.5~24.9 (Normal weight)
* Work at least 75% of full-time work

Exclusion criteria:

* Neurological diseases
* Orthopedic disorders
* Other disorders or regular use of medications known to affect physical activity, autonomic nervous system or pain perception

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy participants with or without chronic neck pain, recruited in Taipei.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Five-minute
  Time domain and frequency domain indices

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taiwan, R.O.C., Taipei, Taiwan